CLINICAL TRIAL: NCT06216327
Title: Veteran-Centered Lethal Means Safety Suicide Prevention Intervention (CDA 19-076)
Brief Title: Home Safety Intervention
Acronym: HSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDX 24-001; 1IK2HX002861-01A2 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Firearm Injury; Overdose
Keywords: firearm
MeSH Terms: conditions — Suicide; Drug Overdose

STUDY DESIGN:
Intervention Model Description: This intervention includes a household safety intervention that is delivered by an interventionist with specific training in facilitating lethal means safety discussions, and the provision of no-cost safety devices for medications and firearms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention arm (Experimental): There is a single intervention arm with no comparator for this pilot study
  Interventions: Behavioral: household safety intervention

INTERVENTIONS:
Behavioral: household safety intervention — This intervention includes a household safety intervention that is delivered by an interventionist with specific training in facilitating lethal means safety discussions, and the provision of no-cost safety devices for medications and firearms.

SUMMARY:
Access to lethal methods of self-harm such as firearms and medications increases risk for suicide. As such, VA/DoD guidelines for the care of individuals with elevated suicide risk include recommendations that clinicians deliver interventions to reduce access to lethal methods of suicide among patients who are identified as having elevated suicide risk. However, no interventions have been developed or tested among Veterans with elevated suicide risk. The aim of this study is to pilot test a lethal means safety intervention developed specifically for Veterans who seek care in VHA clinical settings and are identified as having elevated suicide risk.

DETAILED DESCRIPTION:
The investigators will pilot the LMS intervention among up to 50 Veterans to assess feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Encounter at VHA ED or urgent care setting, outpatient mental health, women's health, or primary care

  ->17 years
* Discharged home from the encounter (rather than hospital admission)
* Positive Columbia Screener
* Patient-reported access to self-owned firearms and/or medications

Exclusion Criteria:

* Unable to consent due to cognitive impairment, severity of illness (including psychiatric symptoms), intoxication with drugs and/or alcohol
* Unreliable telephone access
* Unreliable video access (because remote intervention)
* Those currently experiencing unsheltered homelessness
* No mailing address
* Active opioid or stimulant use disorder
* Active alcohol use disorder with daily alcohol consumption

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment | through study completion, an average of one year
  Ability to recruit 30 Veterans in one year
Feasibility of study follow up | approximately 30 days
  >70% follow up
participant intervention satisfaction | day of intervention delivery - day 0; and at 4 weeks
  >70% with score greater than 23 (Client Satisfaction Questionnaire 8). 8 items, each with 4 answer options (1-4) on a Likert Scale. Likert options are different for each item. Score range is 8 to 32.
participant intervention satisfaction | at 4 weeks
  Qualitative evaluation of participant's experiences
Comfort with intervention discussion | day of intervention delivery - day 0; and at 4 weeks
  "How comfortable did you feel engaging in the discussion? " Likert responses: Very uncomfortable Uncomfortable Neither Comfortable Very comfortable
Intervention helpfulness in medication decisions | day of intervention delivery - day 0; and at 4 weeks
  "How helpful was your interaction in making decisions about medication storage and safety?" Likert responses: Not at all Slightly helpful Moderately helpful Very helpful Extremely helpful
Intervention helpfulness in firearm decisions | day of intervention delivery - day 0; and at 4 weeks
  "How helpful was your interaction in making decisions about firearm storage?" Likert responses: Not at all Slightly helpful Moderately helpful Very helpful Extremely helpful
Respectfulness of the intervention | day of intervention delivery - day 0; and at 4 weeks
  "To what extent was this intervention respectful of your values as a firearm owner? Likert responses: Very disrespectful Disrespectful Neither Respectful Very respectful

SECONDARY OUTCOMES:
Institutional Trust | Day of intervention delivery (day 0) and at 4 weeks
  On a scale from 0 to 10, where 10 indicates complete trust and 0 indicates complete distrust (so 5 would indicate that you neither trust, nor distrust), please indicate your level of trust in the VA healthcare system?
Beliefs about importance of secure medication storage when someone is suicidal | Day of intervention delivery (day 0) and at 4 weeks
  "On a scale of 0 to 10, I want to ask you about whether you find the following safety measures to be important. Someone who answers 0 does not consider them to be important at all, while someone who answers 10 considers them to be extremely important." It is important to securely store medications when I or someone in my household has had recent thoughts of suicide. Answer range: 0-10
Beliefs about importance of secure medication storage always | Day of intervention delivery (day 0) and at 4 weeks
  "On a scale of 0 to 10, I want to ask you about whether you find the following safety measures to be important. Someone who answers 0 does not consider them to be important at all, while someone who answers 10 considers them to be extremely important." It is always important to securely store medications even if someone is not at risk for suicide in the home. Answer range: 0-10
Beliefs about importance of secure firearm storage when someone is suicidal | Day of intervention delivery (day 0) and at 4 weeks
  "On a scale of 0 to 10, I want to ask you about whether you find the following safety measures to be important. Someone who answers 0 does not consider them to be important at all, while someone who answers 10 considers them to be extremely important." It is important to securely store firearms when I or someone in my household has had recent thoughts of suicide. Answer range: 0-10
Beliefs about importance of secure firearm storage always | Day of intervention delivery (day 0) and at 4 weeks
  "On a scale of 0 to 10, I want to ask you about whether you find the following safety measures to be important. Someone who answers 0 does not consider them to be important at all, while someone who answers 10 considers them to be extremely important." It is always important to store firearms securely in a locked space, or with a locking device, even if someone is not at risk for suicide in the home. Answer range: 0-10
Beliefs about importance of unloaded firearm storage always | Day of intervention delivery (day 0) and at 4 weeks
  "On a scale of 0 to 10, I want to ask you about whether you find the following safety measures to be important. Someone who answers 0 does not consider them to be important at all, while someone who answers 10 considers them to be extremely important." It is always important to securely store firearms unloaded even if someone is not at risk for suicide in the home. Answer range: 0-10
Firearm storage storage Stage of Change | Day of intervention delivery at visit #1 (day 0); optional visit #2 (1-29 days); optional visit #3 (2-29 days); and at 4 weeks
  One thing some people consider doing to reduce risk of suicide or injury for themselves and others in their household is to securely store all firearms. On a scale from 0 to 10, where 0 is not at all, and 10 is completely, how would you rate your readiness to [make a change] like that? (range 0-10)
Medication storage storage Stage of Change | Day of intervention delivery at visit #1 (day 0); optional visit #2 (1-29 days); optional visit #3 (2-29 days); and at 4 weeks
  One thing some people consider doing to reduce risk of suicide or injury for themselves and others in their household is to securely store all medications. On a scale from 0 to 10, where 0 is not at all, and 10 is completely, how would you rate your readiness to [make a change]? (range 0-10)
Number of firearms in household | Day of intervention delivery (day 0) and at 4 weeks
  Number of firearms in household: Answer range: 0 to 10,000
Medication adherence | at 4 weeks
  "To what extent have you had difficulty remembering to take your medications in the past month?" Likert responses: Never Rarely Sometimes Very Often Always
Change in firearm storage practices | Day of intervention delivery (day 0) and at 4 weeks
  Changes in whether household firearms are present, and whether present firearms are stored securely. Answers:
  Yes, all of them are locked Yes, some of them are locked None of them are locked I'm not sure
Change in medication storage practices | Day of intervention delivery (day 0) and at 4 weeks
  Changes in whether household medication is present, and whether present medication is stored securely. Answer options:
  Yes, all of the medications in my home are locked up Yes, some of the medications in my home are locked up None of the medications in my home are locked up I'm not sure
Keeping firearms for protection | Day of intervention delivery (day 0) and at 4 weeks
  On a scale of 0 to 10, to what extent do you keep your firearms to protect yourself or your loved ones from other people? Someone who answers 0 does not consider themselves to keep firearms for protection, while someone who answers 10 considers that their firearms are absolutely required for protection. Answer range: 0-10
Firearm removal stage of change | Day of intervention delivery at visit #1 (day 0); optional visit #2 (1-29 days); optional visit #3 (2-29 days); and at 4 weeks
  One of the safest things someone can do while they're going through a difficult time is to store their firearms outside of the home with someone they trust. On a scale from 0 to 10, where 0 is not at all, and 10 is completely, how would you rate your readiness to [make a change] like that? Answer range: 0-10
Change in access to firearm storage combination | Day of intervention delivery (day 0) and at 4 weeks
  Changes in who has access to household locking combinations.
  Answer options:
  You Your spouse or partner Children under the age of 18 years Children 18 years of age or older A friend A neighbor Other:__________
Naloxone prescription | at 8 weeks
  Verification of naloxone prescription within the electronic health record (yes/no)
Change in ammunition storage practices | Day of intervention delivery (day 0) and at 4 weeks
  Changes in whether household ammunition is present, and whether present ammunition is stored securely. Answer options: Yes, all of the ammunition is locked Yes, some of the ammunition is locked None of the ammunition is locked I'm not sure No ammunition is in my home
Medication return envelope | at 8 weeks
  Verification of returned medication safety envelope (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Simonetti, MD MPH, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT06216327/ICF_000.pdf